CLINICAL TRIAL: NCT05218148
Title: Phase II Clinical Study of Oxaliplatin Plus S-1 (SOX) Combined With Sintilimab and Trastuzumab Versus SOX Regimen in the Perioperative Treatment of Locally Advanced HER2-positive Gastric or Gastroesophageal Junction (G/GEJ) Adenocarcinoma
Brief Title: SOX Combined With Sintilimab and Trastuzumab Versus SOX Regimen in the Perioperative Treatment of HER2-positive Locally Advanced Gastric Adenocarcinoma
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Aiping Zhou (Unknown)
Responsible Party: Sponsor-Investigator, Aiping Zhou, Chief physician, Chinese Academy of Medical Sciences
Organization: ChineseAMS (Unknown)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NCC-008261
Record Dates: First submitted 2022-01-16; First posted 2022-02-01 (Actual); Last update posted 2022-04-06 (Actual); Status verified 2022-03

CONDITIONS: HER2-positive; Locally Advanced Solid Tumor; Immunotherapy; Sintilimab; S-1; Oxaliplatin; Gastric or Gastroesophageal Junction Adenocarcinoma
MeSH Terms: interventions — sintilimab; Trastuzumab; S 1 (combination); Oxaliplatin

STUDY DESIGN:
Intervention Model Description: This is an open-label, randomized controlled, exploratory phase II study. Patients with HER2-positive locally advanced gastric or gastroesophageal junction adenocarcinoma who have not received any anti-tumor therapy were randomized in a 1:1 ratio to receive preoperatively: Group A: SOX regimen (oxaliplatin + Seggio) ) + sintilimab + trastuzumab; group B: SOX regimen, 3 cycles of treatment, followed by D2 radical resection, and 5 cycles of adjuvant chemotherapy with the original regimen after surgery
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (Experimental): Group A: SOX regimen (oxaliplatin + Seggio) ) + sintilimab + trastuzumab; 3 cycles of treatment, followed by D2 radical resection, and 5 cycles of adjuvant chemotherapy with the original regimen after surgery
  Interventions: Drug: sintilimab; Drug: Trastuzumab; Drug: S-1 plus oxaliplatin
- Group B (Active Comparator): Group B: SOX regimen, 3 cycles of treatment, followed by D2 radical resection, and 5 cycles of adjuvant chemotherapy with the original regimen after surgery
  Interventions: Drug: S-1 plus oxaliplatin

INTERVENTIONS:
Drug: sintilimab — Sintilimab 200mg was administered as a 30-60 min intravenous (IV) infusion every 3 weeks.3 cycles before surgery and 5 cycles after surgery.
  Arms: Group A
Drug: Trastuzumab — Trastuzumab was 8mg/kg for the first time, and 6mg/kg for the follow-up. 3 cycles before surgery and 5 cycles after surgery.
  Arms: Group A
Drug: S-1 plus oxaliplatin — Oxaliplatin 130 mg/m2 was administered IV every 3 weeks. S-1 was given orally twice daily for the first 2 weeks of each 3-week cycle. The S-1 dose was 40 mg for body surface area (BSA) < 1.25 m2, 50 mg for BSA 1.25 to <1.5 m2 and 60 mg for BSA ≥1.5 m2.
  Body surface area <1.25m2: Tegio 40mg bid day 1 ~ 14; Body surface area 1.25 ~ <1.5m2: Tegio 50mg bid day 1 ~ 14; Body surface area ≥1.5m2: Tegio 60mg bid day 1 ~ 14; 3 cycles before surgery and 3 cycles after surgery.

SUMMARY:
The SOX regimen has became the standard perioperative chemotherapy for locally advanced gastric cancer; The immune checkpoint inhibitors have become a standard treatment for advanced or metastatic gastric cancer；For HER2-positive locally advanced gastric cancer, some phase II studies have shown that chemotherapy combined with trastuzumab can further improve the pathological remission rate;This prospective phase II clinical trial was designed, using SOX combined with sintilimab and trastuzumab to treat HER2 positive locally advanced gastric or gastroesophageal junction adenocarcinoma patients.

DETAILED DESCRIPTION:
This phase II trial is a single-arm and single-center clinical study. Neoadjuvant chemotherapy is a standard treatment for locally advanced gastric cancer. The SOX regimen has became the standard perioperative chemotherapy regimen for locally advanced gastric cancer. For HER2-positive locally advanced gastric cancer, the neoadjuvant treatment is still based on chemotherapy alone. Some phase II studies have shown that chemotherapy combined with trastuzumab can further improve the pathological response. But it has not yet become a standard treatment strategy.

In the field of gastric cancer, checkpoint inhibitors have become a standard treatment for advanced or metastatic gastric cancer. PD-1 monoclonal antibody (Sintilimab) + trastuzumab + chemotherapy (SOX regimen ) may be an ideal perioperative treatment for HER2-positive locally advanced gastric cancer.

ELIGIBILITY:
Inclusion Criteria:

* Sign the informed consent form.
* Locally advanced adenocarcinoma of the stomach or gastroesophageal junction (Siewert type II/III) confirmed by pathology or cytology.
* The definition of a positive HER2 test result is as follows: IHC detects HER2 3+ or IHC detects HER2 2+ and FISH is positive.
* Clinically, based on chest, abdomen and pelvic CT, gastroscopy, endoscopic ultrasonography, gastrointestinal contrast, ordinary ultrasound, or laparoscopy if possible, it is judged as T3-4a N+ or T4bN any gastric cancer or gastroesophageal junction cancer (refer to AJCC Article Version 8 in stages).
* Patients have not received chemotherapy and/or immunotherapy and/or trastuzumab treatment and/or radiotherapy in the past.
* Age 18-75 years old.
* The Eastern Cooperative Oncology Group (ECOG) performance status score was 0 or 1, and there was no deterioration within 2 weeks before the first administration of the study drug.
* Good organ function:

Blood routine: hemoglobin ≥90g/L, white blood cell ≥3.0×109/L, neutrophil ≥1.5×109/L, platelet ≥100×109/L; Renal function: creatinine≤1.5×upper limit of normal (UNL) or creatinine clearance ≥60ml/min; Liver function: total bilirubin (TBIL)≤1.5×upper limit of normal (UNL); ALT≤2.5×UNL, AST≤2.5×UNL.

Exclusion Criteria:

* The pathology is other types besides adenocarcinoma, such as squamous cell carcinoma, adenosquamous carcinoma, neuroendocrine carcinoma and so on.
* Have received chemotherapy and/or radiotherapy in the past.
* Have received any anti-PD-1, anti-PD-L1/L2 antibodies, anti-CTLA-4 antibodies and other immunotherapy in the past.
* Have received any anti-HER2 therapy in the past.
* Intra-abdominal dissemination or distant metastasis (M1).
* Clinically significant ascites.
* Known to have allergic reactions to oxaliplatin and any ingredients or excipients of Tiggio.
* Known to have allergic reactions to any ingredients or excipients of Sintilimab and Trastuzumab.
* Inability to swallow, intestinal obstruction, or other factors that affect the administration and absorption of the drug.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Estimated)
Dates: Start 2022-04-01 (Estimated); Primary Completion 2024-10-01 (Estimated); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
Major pathological response rate (MPR) | Up to 6 months
  Proportion of subjects with residual tumor less than 10% or complete response

SECONDARY OUTCOMES:
Pathological response rate (refer to Becker-TRG evaluation standard) | Up to 3 years
  TRG level 1-3:
  1a: No tumor remains at all
  1b: Less than 10% of the tumor remains 2: 10%-50% tumor residual 3: More than 50% of the tumor remains or there is no change in the tumor
Objective response rate (ORR) | Up to 3 years
  Proportion of subjects with initial RECIST 1.1 measurable disease who have complete response (CR) or partial response (PR) according to iRECIST
Disease-free survival (DFS) | Up to 3 years
  Time from Cycle 1 Day 1 treatment administration to the first documented event of: disease progression, disease recurrence following surgery (preferably biopsy proven), or death - whichever occurs first.
Overall survival (OS) | Up to 3 years
  Time from Cycle 1 Day 1 treatment administration to death due to any cause.
Incicende of Adverse Events (AEs) | Up to3 years
  Number of patients with AE, treatment-related AE (TRAE), immune-related AEs (irAE), AE of special interest (AESI), serious adverse event (SAE) assessed by CTCAE v5.0.
Biomarker assessment | Up to3 years
  To analyze the differences of gene and immune microenvironment biomarkers among patients with different curative effects, and further explore the relationship with the efficacy of clinical treatment.
  To analyze the correlation between peripheral blood indexes and the efficacy of clinical treatment.

CONTACTS AND LOCATIONS:
Locations (1):
- Cancer Hospital & Institute, Chinese Academy of Medical Sciences, Beijing, China

IPD SHARING:
Plan to Share IPD: No